CLINICAL TRIAL: NCT00704652
Title: Evaluation of Functional and Morphological Retinal Changes in the Course of Systemic Aranesp Treatment in Patients With Diabetes Mellitus
Brief Title: Evaluation of Retinal Changes in Systemic Darbepoetin Alpha Treatment in Patients With Diabetes Mellitus
Acronym: EPOinDR
Status: Terminated | Type: Observational
Why Stopped: Patient recruitment was not sufficient to achieve the needed patient numbers.
Sponsor: Medical University of Vienna (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Gabor Deak, MD, Medical University of Vienna
Other Study IDs: 394/2007
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Diabetic patients suffering from renal insufficiency with stable haemoglobin levels (receiving no EPO supplementation)
- B: Diabetic patients with renal insufficiency and in need of recombinant human EPO (darbepoetin alfa) substitution because of inadequate erythropoiesis. In both groups the target haemoglobin level is 10-12 gHb/ml, all treatment is performed according to label.

SUMMARY:
The purpose of this study is to determine whether systemic administration of darbepoetin alpha results in the progression or regression of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Males and females aged 18 to 80 yrs
* Diabetes mellitus type 1 or 2
* Haemoglobin level above the treatment threshold level (as described in the drug description)
* Receiving no darbepoetin alfa treatment
* Best Corrected Visual Acuity (BCVA) better than 20/200
* No clinically significant macular edema (CSME) or CSME already treated with laser photocoagulation.

Group B:

* Males and females aged 18 to 80 yrs
* Diabetes mellitus type 1 or2
* Anaemia (due to renal failure), haemoglobin level under the treatment threshold level before the initialisation of the therapy (as described in the drug label)
* Starting to receive darbepoetin alfa treatment (darbepoetin alfa, Aranesp, Amgen)
* BCVA better than 20/200
* No clinically significant macular edema (CSME) or CSME already treated with laser photocoagulation.

Exclusion Criteria:

* History of retinal disease other than DR
* History of intraocular surgery, including laser treatment in the past 4 month
* A major change in the insulin treatment of the patient in the past 4 month or during the follow up period.
* Inability to communicate in German or English
* Dementia; inability to follow commands
* Epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with min. Grade 2 renal insufficiency, and in Group B with anemia that is to be treated with systemic ESA therapy.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Morphologic changes in the retina detected by HD-OCT following darbepoetin alpha therapy compared to control patients | 9 month

SECONDARY OUTCOMES:
Functional improvement in best corrected visual acuity (BCVA) and microperimetry following darbepoetin alpha therapy compared to control patients. | 9 month
Changes in anterior chamber flare and cell count following darbepoetin alpha therapy compared to control patients. | 9 month
Changes in the fundus image and fluorescein angiographic features following darbepoetin alpha therapy compared to control patients. | 9 month
Changes in blood count, chemistry, Astrup and blood clotting following darbepoetin alpha therapy compared to control patients. | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, Prof., Principal Investigator — Departmen of Ophthalmology, Medical Unversity of Vienna
Locations (1):
- Departmen of Ophthalmology, Medical Unversity of Vienna, Vienna, Vienna, Austria